CLINICAL TRIAL: NCT03210194
Title: Continuous Training and Certification in Neonatal Resuscitation in Remote Areas Using a Multi-platform Information and Communication Technology Intervention Compared to Standard Training: A Randomized Cluster Trial
Brief Title: Randomized Cluster Trial on Innovative and Standard Strategies for Neonatal Resuscitation Training (RCPNEOPERU Project)
Acronym: RCPNEOPERU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Grand Challenges Canada (Other); Instituto Nacional de Salud del Niño. Lima, Peru (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 100651
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Neonatal Asphyxia
Keywords: Inservice Training; Neonatal Resuscitation; Randomized Cluster Trial
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Neonatal Resuscitation Training (Active Comparator): Standard training will be conducted through a theoretical-practical course, which will be administered once during the study period, to all health professionals of the selected facilities, according to the randomization. It is an 8-hour course, with 3 hours of theory and 5 hours of practice, which will take place during a single day. The course will be performed by staff of the Neonatal Unit of the Instituto Nacional de Salud del Niño (National Institute of Child Health, Lima, Peru), and will be coordinated by an NRP instructor accredited by the American Academy of Pediatrics. Participants who have completed their attendance to theoretical sessions, participated in the simulated practices and approved the printed exams taken the same day will we granted a Standard Certification.
  Interventions: Behavioral: Standard Neonatal Resuscitation Training
- MP-ICT Neonatal Resuscitation Training (Experimental): The Multi-platform ICT (MP-ICT) training includes continuous certification in neonatal resuscitation and is being developed for online and offline access, and will be complemented with simulated practices on every site. The platform is being improved and adjusted to the needs of the fieldwork in Ayacucho and Cusco. The adaptations include increasing hosting; ameliorate friendly usability, uploading packages and videos, improvement of examination and certifications, and tests for readiness. The MP-ICT resource will be accessed from remote Peruvian locations through computers, personal portable devices and cell phones. To be granted an MP-ICT Certification the trainee needs to have passed the online theoretical exam, assist to the practice and approve practical skills assessment.
  Interventions: Behavioral: MP-ICT Neonatal Resuscitation Training

INTERVENTIONS:
Behavioral: Standard Neonatal Resuscitation Training — Theoretical and practical training on basic and advanced neonatal resuscitation skills, directed to personnel from remote health centers using Standard Training
  Other Names: Standard Training
  Arms: Standard Neonatal Resuscitation Training
Behavioral: MP-ICT Neonatal Resuscitation Training — Theoretical and practical training on basic and advanced neonatal resuscitation skills, directed to personnel from remote health centers using Information and Communication Technologies
  Other Names: Multi-platform ICT training (MP-ICT)
  Arms: MP-ICT Neonatal Resuscitation Training

SUMMARY:
Background: About 10% of all newborns may have difficulty breathing and require support by trained personnel. In Peru, 90% of deliveries occur in health facilities; however there is not a national neonatal resuscitation and certification program for the public health sector. In addition, the Andes and the Amazon regions concentrate large rural remote areas, which further limit the implementation of training programs and the accomplishment of continuous certification. Neonatal resuscitation training through the use of information, communication and technology (ICT) tools running on a computer, tablet or mobile phone may overcome such limitations. This strategy allows online and offline access to educational resources, paving the way to more frequent and efficient training and certification processes.

Objective: To evaluate the effects of a neonatal resuscitation training and certification program that uses a multi-platform ICT (MP-ICT) strategy on neonatal health care in remote areas.

Methods: The investigators propose to conduct the study through a cluster-randomized trial, where the study and analysis units are the health care facility. Eligible facilities will include primary and secondary health care level facilities that are located in provinces with neonatal mortality rates higher than 15 per 1,000 live births. The investigators will compare the proportion of newborns with a heart rate ≥100 beats per minute at 2 minutes after birth in health care facilities that receive MP-ICT training and certification implementation, with those that receive conventional training and certification.

Discussion: The investigators expect that the intervention show to be more effective than the current standard of care. The investigators are prepared to include it within a national neonatal resuscitation training and certification program to be implemented at national scale together with policymakers and other key stakeholders.

DETAILED DESCRIPTION:
Background

A training system using Multi-platform ICT (MP-ICT) tools offers reliable and easier access to information and training packages from different locations which can be implemented even in rural settings without access to internet. Platforms may be available online, and users can download the training content through a personal computer, a tablet or a mobile phone. The training content may be downloaded repeatedly afterwards, even in remote areas without access to internet.

Our project aims to evaluate the performance of a continuous process of training and certification in neonatal resuscitation in primary and secondary health facilities in the departments of Ayacucho and Cusco, through the use of MP-ICT tools. It aims at providing proof of concept of the interventions, which then could be expected to be incorporated as a component of a national neonatal resuscitation program to be implemented nationwide.

The traditional way to train and certify health care professionals is through administration of a theoretical expositive course, reinforced subsequently by a practical component. This modality requires face-to-face contact between trainers and trainees. Health workers need to move from their job site to the instruction sites, usually located in the capital city of the department or in the capital city of the country. This poses economic and logistic challenges to both health authorities and health workers, and results in erratic frequency and low uptake of training courses.

Research hypothesis

The use of multi-platform ICT strategies for training and certification in neonatal resuscitation will increase the proportion of children with heart rate equal or greater than 100/minute at two minutes of life, as compared to standard training.

Primary objective

To evaluate the effects of the use of a Multi-Platform ICT strategies for training and certification on neonatal resuscitation in first and second level health facilities of Ayacucho and Cusco departments.

Settings

Ayacucho and Cusco are two Peruvian regions located to the south of the country. These regions cover areas of Andean highlands, but their territory is mainly on the Amazon rainforest. Also, in those departments there is the "Valley of the Apurímac, Ene and Mantaro Rivers", also known as the VRAEM, which is a geopolitical extremely poor area and one of the major areas of coca growing in Peru.

According to Peruvian Registry of Institutions that Provide Health Services (RENIPRESS), Ayacucho has 418 and Cusco 848 registered health facilities.

Study design

The proposed study design is a randomized cluster trial. The Units of study and analysis will be first and second level health facilities from Ayacucho and Cusco departments. Each health facility will be a cluster. Clusters will be randomly assigned either to the MP-ICT course and certification package (intervention) or to the standard training and certification package (control).

Sample size

The investigators would require 12 clusters (health facilities), divided in 6 clusters for each one of two arms, and with an average of 334 deliveries per facility in the observation period.

Assuming the occurrence of about 4,000 births during a period of 6 months of filed study observation, the investigators aim at discriminating a 4% difference in the proportion of newborns with heart rate equal or greater 100 beats per minute at 2 minutes of life between the intervention and the control group. The proposed power of study is 80% and the acceptable alpha error is 5%. The percentage for heart rate >100 bpm at 2 minutes of life, during suitable resuscitation using self-inflated bag is 90% and it is the expected value for the intervention group. For the control group it is expected at least 4 points below the value achieved in the intervention group (i.e. no more than 86%).

Description of interventions

Standard Training

Standard training will be conducted through a theoretical-practical course, which will be administered once during the study period, to all health professionals of the selected facilities, according to the randomization. It is an 8-hour course, with 3 hours of theory (based on suggested readings) and 5 hours of practice, which will take place during a single day, approximately from 9:00 a.m. to 6:00 p.m according to the availability of the trained instructors and participants on suitable facilities for skills training. The course will be performed by staff of the Neonatal Unit of the Instituto Nacional de Salud del Niño (National Institute of Child Health, Lima, Peru), and will be coordinated by an Neonatal Resuscitation Program (NRP) instructor accredited by the American Academy of Pediatrics.

Participants who have completed their attendance to theoretical sessions, participated in the simulated practices and approved the printed exams taken the same day will grant a Standard Certification. The practice will be evaluated qualitatively in terms of assistance, participation and performance of activities.

Multi-platform ICT training

The continuous process of training and certification in neonatal resuscitation will be developed as a multi-platform format, including theory rechargeable online and accessible offline, and will be complemented with simulated practices. The Practical Component will be made after the Theoretical one and the activities will be completed according to the availability of the trained instructors and participants on suitable facilities for skills training.

The platform contains training packages, and links to review and download neonatal resuscitation tools, technical documents, and regulatory information. During the first three months of the project the platform is being improved and adjusted to the needs of the fieldwork in Ayacucho and Cusco. The adaptations include increasing hosting; ameliorate friendly usability, uploading packages and videos, improvement of examination and certifications, and tests for readiness. The MP-ICT resource will be user-friendly and can be accessed from remote locations through computers, personal portable devices and cell phones. It allows downloading of the different documents, and that facilitates learning and evaluation in an interactive and virtual way, without the physical presence of instructors or teachers. However, through the website the investigators can generate virtual meetings as forums or chat. In addition, the website will allow the programming of simulated practices, with the presence of the instructor.

Authorized participants will be able to download the information for the theoretical activities in 4 packages: Package A, B, C and D: each one containing interactive tools as videos-360 and action mazes (as Quandary), and other videos, documents or short text to read in Spanish. After downloading this information, the tests are enabled in sequence: When approve part A and B, it will be enable part C and D. The interactivity is expressed in 360º videos allowing the user to change the observation point in a recorded environment. The interactivity for action mazes (like Quandary) has demonstrated that feedback-oriented interactive exercises increase higher-order cognitive skills.

To be granted an MP-ICT Certification the trainee needs to have passed the online theoretical exam, assist to the practice and approve practical skills assessment.

Randomization

Computer-generated random numbers will be used to assign the selected health facilities to either MP-ICT training (Intervention Group) or to standard training (Control Group). There will be a matching process of health facilities by proportion of groups of non-medical professionals (nurses and obstetricians) and by availability of basic equipment and maternal and newborn care supplies, to ensure that health facilities are comparable. Once paired, they will be randomly allocated through a blocked randomization, to ensure a balanced distribution of facilities in each group.

Effectiveness assessment

After randomization of each facility, standard training or MP-ICT training will be conducted. Evaluations will include a baseline assessment of available equipment and supplies for neonatal resuscitation, immediately after enrolment and before training. To determine the duration of the effects of the intervention, the proposed outcome indicators will be evaluated six months after the training. The primary and secondary outcomes will be assessed intrapartum (within 5 minutes after birth) and postpartum (at 24 hours and 7 days, to know the outcome of the infant). The assessments will be based on an observation sheet, in which trained research assistants (registered nurses or equivalent local personnel) will record the activities conducted during the delivery and the birth, and the results of the neonatal resuscitation. The observation of performance in neonatal resuscitation can also be recorded randomly through videos, to verify the validity of the data collected by the research assistant. The videos will be reviewed by the field monitor and by one of the investigators. In order to comply with confidentiality requirements, the videos will be deleted after verification of information.

Statistical analysis

An intention to treat analysis will be performed, including all clusters as they were initially assigned, including premature withdrawals. Additionally, a per-protocol analysis will be carried out, where only clusters that have completed the study protocol will be considered. The primary outcome will be compared in each arm using chi-square if the variable of distribution is normal, or alternatively through the Fisher's exact test. Secondary outcomes will be compared using the Student's t-test or the Kruskal-Wallis test, the chi-square test or Fisher's exact test.

Staff training

The investigators will resort to local staff as research assistants including the field supervisor. They will conduct the preparatory work and the study procedures, including information presentations, informed consent administration, observation of case management, and completion of case report forms. Such personnel will be trained in the conduction of studies complying with the standards of good practice, before the study initiation.

Ethical aspects and confidentiality

The proposal, instruments and consent forms have been approved by the Ethics Committee of the Universidad Peruana Cayetano Heredia. Written authorization will be obtained from the authorities of the Regional Health Departments (DIRESAS) involved and from the authorities of the health facilities. Written informed consent will be obtained from the health professionals who will participate in the neonatal resuscitation training. Written informed consent of the mothers will also be obtained for the collection of birth and newborn data.

The information obtained will be codified and personal identification data like names and date of birth will be deleted to protect confidentiality. Data access will be limited to the Principal Investigator and authorized Co-Investigators. The study documents will be stored in locked environments at the Centro de Investigación para el Desarrollo Integral y Sostenible (CIDIS) at Universidad Peruana Cayetano Heredia to which access will be granted only to the Principal Investigator and the Co-Investigators authorized by the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary level facilities located in Ayacucho and Cusco that have a neonatal mortality rate higher than 15 per 1,000 livebirths will be eligible

Exclusion Criteria:

* Health facilities whose authorities refuse participation of their health professionals, facilities with less than 290 births a year, facilities located at more than 210 kilometres from the department capital and those located in high risk areas due to social unrest will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Heart rate at two minutes of life | Up to six months
  Percentage of infants with heart rate equal or greater than 100 per minute at 2 minutes of life.

SECONDARY OUTCOMES:
Starting positive pressure ventilation | Up to six months
  Time to start positive pressure ventilation after birth
Heart rate >= 100 bpm | Up to six months
  Time to achieve heart rate greater or equal than 100 per minute
Apgar | Up to six months
  Apgar at 1 minute and at 5 minutes
Oxygen requirement at 10 minutes | Up to six months
  Use of supplemental oxygen after 10 minutes of life
Oxygen requirement at 30 minutes | Up to six months
  Inspiratory oxygen fraction needed at 30 minutes after birth
Early neonatal mortality | Up to six months
  Mortality rate during the first 7 days of life
Early neonatal referral | Up to six months
  Number of referrals to health facilities with greater resolution capacity during the first 7 days of life
Certified NRP providers | Up to six months
  Number of certified health professionals as providers
Certified NRP instructors | Up to six months
  Number of certified health professionals as instructors

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Delgado, PhD, Principal Investigator — Universidad Nacional Mayor de San Marcos, School of Medicine, Department of Pediatrics, NEO research group; Instituto Nacional de Salud del Niño, Neonatal Unit; Universidad Peruana Cayetano Heredia, CIDIS and MAMAWAWA research centers. Lima-Peru
Locations (1):
- Instituto Nacional de Salud del Niño, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] Lawn JE, Kerber K, Enweronu-Laryea C, Cousens S. 3.6 million neonatal deaths--what is progressing and what is not? Semin Perinatol. 2010 Dec;34(6):371-86. doi: 10.1053/j.semperi.2010.09.011. PMID 21094412
- [Background] Huicho L, Canseco FD, Lema C, Miranda JJ, Lescano AG. [Incentives to attract and retain the health workforce in rural areas of Peru: a qualitative study]. Cad Saude Publica. 2012 Apr;28(4):729-39. doi: 10.1590/s0102-311x2012000400012. Spanish. PMID 22488318
- [Background] Huicho L, Segura ER, Huayanay-Espinoza CA, de Guzman JN, Restrepo-Mendez MC, Tam Y, Barros AJ, Victora CG; Peru Countdown Country Case Study Working Group. Child health and nutrition in Peru within an antipoverty political agenda: a Countdown to 2015 country case study. Lancet Glob Health. 2016 Jun;4(6):e414-26. doi: 10.1016/S2214-109X(16)00085-1. PMID 27198845
- [Background] Huicho L, Huayanay-Espinoza CA, Herrera-Perez E, Nino de Guzman J, Rivera-Ch M, Restrepo-Mendez MC, Barros AJ. Examining national and district-level trends in neonatal health in Peru through an equity lens: a success story driven by political will and societal advocacy. BMC Public Health. 2016 Sep 12;16 Suppl 2(Suppl 2):796. doi: 10.1186/s12889-016-3405-2. PMID 27634453
- [Background] Avila J, Tavera M, Carrasco M. [Epidemiological characteristics of neonatal mortality in Peru, 2011-2012]. Rev Peru Med Exp Salud Publica. 2015 Jul-Sep;32(3):423-30. Spanish. PMID 26580922
- [Background] Perlman J, Kattwinkel J, Wyllie J, Guinsburg R, Velaphi S; Nalini Singhal for the Neonatal ILCOR Task Force Group. Neonatal resuscitation: in pursuit of evidence gaps in knowledge. Resuscitation. 2012 May;83(5):545-50. doi: 10.1016/j.resuscitation.2012.01.003. Epub 2012 Jan 13. PMID 22245921
- [Background] Niermeyer S. From the Neonatal Resuscitation Program to Helping Babies Breathe: Global impact of educational programs in neonatal resuscitation. Semin Fetal Neonatal Med. 2015 Oct;20(5):300-8. doi: 10.1016/j.siny.2015.06.005. Epub 2015 Aug 8. PMID 26265602
- [Background] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Background] Elsensohn AN, Ricks DJ, Ota A, Nevers SW, Channell N, Liaqat M, Ricks JH, Villanueva AM. The success of Peru's Neonatal Resuscitation Initiative. Arch Dis Child Fetal Neonatal Ed. 2013 Jul;98(4):F375-6. doi: 10.1136/archdischild-2013-303864. Epub 2013 May 18. No abstract available. PMID 23685438
- [Background] Huicho L, Trelles M, Gonzales F, Mendoza W, Miranda J. Mortality profiles in a country facing epidemiological transition: an analysis of registered data. BMC Public Health. 2009 Feb 2;9:47. doi: 10.1186/1471-2458-9-47. PMID 19187553
- [Derived] Delgado CA, Gomez Pomar EM, Velasquez P, Sanchez V, Shimabuku R, Huicho L; RCPNEOPERU Study Group. Continuous training and certification in neonatal resuscitation in remote areas using a multi-platform information and communication technology intervention, compared to standard training: A randomized cluster trial study protocol. F1000Res. 2017 Aug 30;6:1599. doi: 10.12688/f1000research.12269.3. eCollection 2017. PMID 30026911